CLINICAL TRIAL: NCT05006820
Title: Epidemiology of Roller Hockey Related Injuries.
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Hugo Olmedillas Fernandez, Associate professor, University of Oviedo
Other Study IDs: UO2021-02
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Sports Injury
Keywords: Prevalence; Multidirectional Sport; Injury prevention; Athletic injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No intervention

SUMMARY:
Roller Hockey is a sport played on a 40*20 metres rink characterized by combined periods of high intensity and short breaks, there´s a lack of epidemiological studies in this field. In line with the well-established model of sports injury prevention research proffered by van Mechelen, the first stage in this process is establishing the extent of the problem i.e. injury incidence, severity and burden. Through an online survey filled by semiprofessional athletes, it is posible to obtain all this important information. This way, it will be possible to fulfill a gap in the literature and take action in the near future in order to reduce the prevalence of injuries in this sport.

DETAILED DESCRIPTION:
A retrospective study was performed in male Roller Hockey players. 275 players will be recruited. Data of all injury along a whole season will be collected. Patients' information, including age, number of years playing, skill level and injured body part, will be analysed.

ELIGIBILITY:
Inclusion Criteria: Being a roller hockey player, play for one of the teams who participated in the 2020-2021 season third division league (Ok Liga Bronce). Play in at least one match in the season.

-

Exclusion Criteria: Being unable to understand the questionaire, do not accept on participating in the study.

-

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Roller Hockey players playing in the spanish senior´s third division league
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Injury prevalence | September 2020-June 2021
  Injury prevalence rates [Injury prevalence rates calculated per 1000 hours of play]

SECONDARY OUTCOMES:
Injury burden | September 2020-June 2021
  Days lost per 1000 hours of exposure
Injury prevalence according to occurrence | September 2020-June 2021
  Number of injuries sustained during training/ Number of injuries sustained during a match (% of all)
Injury prevalence by mechanism of injury | September 2020-June 2021
  Number of injuries according to the mechanism of injury (Contact (Direct or indirect) or Non-Contact) (% of all)
Injury prevalence according to location | September 2020-June 2021
  Distribution of injuries according to location of the injury (on the body, % of all)
Injury prevalence according to tissue affected | September 2020-June 2021
  Description of the distribution of injuries according to the type of the injury (muscle only) (% of all)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Olmedillas, PhD, Principal Investigator — Universidad de Oviedo
Locations (1):
- Hugo Olmedillas, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No